CLINICAL TRIAL: NCT01686204
Title: Reduction of Obesity-Associated Intestinal Inflammation by Low-Fat Dairy Yogurt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Dairy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-0669
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Intestinal Barrier Function; Chronic Inflammation
Keywords: Yogurt; Intestine; Inflammation; Obese
MeSH Terms: conditions — Inflammation; Obesity

ARMS (2):
- Non-obese individuals (Active Comparator): Daily consumption of 12 oz lowfat yogurt or soy pudding for 9 weeks.
  Interventions: Other: Low fat dairy yogurt; Other: Soy pudding
- Obese individuals (Experimental): Consumption of 12 oz of soy pudding or low fat dairy yogurt daily for 9 weeks.
  Interventions: Other: Low fat dairy yogurt; Other: Soy pudding

INTERVENTIONS:
Other: Low fat dairy yogurt — Consumption of 12 oz of low fat dairy yogurt daily for 9 weeks
Other: Soy pudding — Consumption of 12 oz of low fat soy pudding daily for 9 weeks.

SUMMARY:
The main objective of this work is to conduct a clinical trial in obese and non-obese individuals testing the ability of low-fat dairy yogurt to improve gastrointestinal health and reduce chronic inflammation. Our central hypothesis is that short and long-term consumption of low-fat dairy yogurt will reduce inflammation to a greater extent in obese individuals by improving intestinal barrier function.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women
* BMI from 18.5-27 and 30-40 kg/m2
* resting blood pressure <140/90 mmHg
* not taking medication to control hypertension
* stable body weight for the previous 2 months
* willing to maintain a normal exercise level and avoid exercise 24 h prior to blood sampling
* willing to avoid yogurt and probiotic-containing foods or consume 2 servings of yogurt for the duration of the study

Exclusion Criteria:

* previous diagnoses of cardiovascular disease (CVD), diabetes, or arthritis (except for osteo-arthritis)
* currently being treated for cancer (i.e., chemotherapy, radiation therapy)
* prescribed estrogen replacement therapy
* practicing weight-loss, vegetarian, kosher, or vegan diets
* currently taking dietary supplements
* exceed alcohol consumption more than moderate drinking (1 drink/day or a total of 7/week)
* actively using antibiotics
* taking anti-inflammatory drugs
* have allergies to soy, egg or milk
* perimenopausal or menopausal symptoms

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09-30 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Plasma soluble cluster of differentiation 14 (sCD14) | 0, 3, 6, and 9 wk
  Fasting plasma sCD14 (change from baseline)

SECONDARY OUTCOMES:
Fasting plasma interleukin-6 (IL-6) | 0, 3, 6, 9 wk
  Fasting plasma IL-6 (change from baseline)
Postprandial sCD14 | 0 and 9 wk
  Postprandial plasma sCD14 following a high-fat, high-calorie challenge meal (area under curve)
Postprandial interleukin-6 (IL-6) | 0 and 9 wk
  Postprandial plasma IL-6 following a high-fat, high-calorie challenge meal (area under curve)

OTHER OUTCOMES:
Fasting lipopolysaccharide binding protein (LBP) | 0 and 9 wk
  Determined by immunoassay
Fasting plasma endotoxin (LPS, lipopolysaccharide) | 0, 9 wk
  Determined by limulus amebocyte lysate assay
Fasting plasma core antibodies to endotoxin | 0 and 9 wk
  Immunoglobulin M Endotoxin-core antibody (IgM EndoCAb)
Fasting plasma anandamide (AEA) | 0, 9 wk
  Determined by LC-MS
Fasting plasma 2-arachidonoylglycerol (2-AG) | 0, 9 wk
  Determined by LC-MS
Fasting plasma IL-10 | 0, 9 wk
  Determined by immunoassay
Fasting plasma high-sensitivity C-reactive protein (hsCRP) | 0, 9 wk
  Determined in fasting plasma
Fasting plasma Tumor Necrosis Factor-alpha (TNF-α) | 0, 9 wk
  Determined in fasting plasma
Fasting plasma Soluble TNF-Receptor II (sTNF-RII) | 0, 9 wk
  Determined in fasting plasma
TNF-alpha/sTNF-RII ratio | 0, 9 wk
  Determined in fasting plasma
Fasting plasma glucose | 0, 9 wk
  Determined in fasting plasma
Fasting plasma triglycerides | 0, 9 wk
  Determined in fasting plasma
Fasting plasma insulin | 0, 9 wk
  Determined in fasting plasma
Fasting plasma soluble cluster of differentiation 14 (sCD14) | 0, 9 wk
  Determined in fasting plasma
Body weight | 0, 3, 6, 9 wk
Body mass index | 0, 3, 6, 9 wk
Waist circumference | 0, 3, 6, 9 wk
Systolic blood pressure | 0, 3, 6, 9 wk
Diastolic blood pressure | 0, 3, 6, 9 wk
Fasting RPLP0, encoding ribosomal protein large P0 | 0, 9 wk
  mRNA expression of peripheral blood mononuclear cell normalized to encoding 18s rRNA (RNA18S5)
TLR4, encoding Toll-like receptor 4 | 0, 9 wk
  mRNA expression of peripheral blood mononuclear cell normalized to encoding 18s rRNA (RNA18S5)
RELA, encoding p65 subunit of nuclear factor kappa B | 0, 9 wk
  mRNA expression of peripheral blood mononuclear cell normalized to encoding 18s rRNA (RNA18S5)
NFKBIA, encoding nuclear factor kappa B inhibitor alpha | 0, 9 wk
  mRNA expression of peripheral blood mononuclear cell normalized to encoding 18s rRNA (RNA18S5)
PTGS2, encoding cyclooxygenase-2 (COX-2) | 0, 9 wk
  mRNA expression of peripheral blood mononuclear cell normalized to encoding 18s rRNA (RNA18S5)
NCF1,encoding the p47 subunit of nicotinamide adenine dinucleotide phosphate-oxidase, (NADPH oxidase) | 0, 9 wk
  mRNA expression of peripheral blood mononuclear cell normalized to encoding 18s rRNA (RNA18S5)
TNF, encoding tumor necrosis factors (TNF) | 0, 9 wk
  mRNA expression of peripheral blood mononuclear cell normalized to encoding 18s rRNA (RNA18S5)
IFNG, encoding interferon-γ | 0, 9 wk
  mRNA expression of peripheral blood mononuclear cell normalized to encoding 18s rRNA (RNA18S5)
TGFB1, encoding transforming growth factor beta 1 (TGFβ1) | 0, 9 wk
  mRNA expression of peripheral blood mononuclear cell normalized to encoding 18s rRNA (RNA18S5)
Postprandial plasma glucose | 0, 9 wk
  Postprandial plasma glucose following a high-fat, high-calorie challenge meal (area under curve)
Postprandial plasma triglycerides | 0, 9 wk
  Postprandial plasma triglycerides following a high-fat, high-calorie challenge meal (area under curve)
Postprandial lipopolysaccharide binding protein (LBP) | 0, 9 wk
  Postprandial plasma LBP following a high-fat, high-calorie challenge meal (area under curve)
Postprandial lipopolysaccharide (LPS) | 0, 9 wk
  Postprandial plasma LPS following a high-fat, high-calorie challenge meal determined by limulus amebocyte lysate assay (area under curve)
Postprandial lipopolysaccharide binding protein (LBP)/soluble cluster of differentiation 14 (sCD14) ratio | 0, 9 wk
  Postprandial LBP/sCD14 ratio following a high-fat, high-calorie challenge meal (area under curve)
Postprandial plasma insulin | 0, 9 wk
  Postprandial plasma insulin following a high-fat, high-calorie challenge meal (area under curve)
Energy intake (kcal) | 0, 9 wk
  Self-reported food intake determined by dietary records
Total fat (g) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Carbohydrate (g) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Total protein (g) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Total fat (%) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Carbohydrate (%) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Total protein (%) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Cholestrol (mg) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Saturated fatty acids (g) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Vitamin D (μg) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Calcium (mg) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Sodium (mg) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Potassium (mg) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Total sugars (g) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records
Added sugars (g) | 0, 9 wk
  Self-reported nutrient intake determined by dietary records

CONTACTS AND LOCATIONS:
Overall Officials: Bradley W Bolling, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Department of Food Science, Babcock Hall, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Pei R, DiMarco DM, Putt KK, Martin DA, Chitchumroonchokchai C, Bruno RS, Bolling BW. Premeal Low-Fat Yogurt Consumption Reduces Postprandial Inflammation and Markers of Endotoxin Exposure in Healthy Premenopausal Women in a Randomized Controlled Trial. J Nutr. 2018 Jun 1;148(6):910-916. doi: 10.1093/jn/nxy046. PMID 29767743
- [Derived] Pei R, DiMarco DM, Putt KK, Martin DA, Gu Q, Chitchumroonchokchai C, White HM, Scarlett CO, Bruno RS, Bolling BW. Low-fat yogurt consumption reduces biomarkers of chronic inflammation and inhibits markers of endotoxin exposure in healthy premenopausal women: a randomised controlled trial. Br J Nutr. 2017 Dec;118(12):1043-1051. doi: 10.1017/S0007114517003038. Epub 2017 Nov 28. PMID 29179781